CLINICAL TRIAL: NCT03909945
Title: Rationale and Design of a Single Arm, Non-randomized Open-label Clinical Trial Evaluating a Tablet Made of Aqueous Extract of Annona Muricata in an African Hypertensive Population
Brief Title: Evaluation of an Antihypertensive Food Supplement Based on Aqueous Extract From Annona Muricata Sheets
Acronym: AM-HTN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANNOMUPRIL
Record Dates: First submitted 2019-03-05; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Hypertension
Keywords: Annona muricata; Hypertension; Sub saharan Africa
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Before and after study intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): The intervention consisted in the daily administration, during 60 days, of a 796 mg tablet of aqueous extracts of leaves of Annona muricata between 08:00 AM and 09:00 AM.
  Interventions: Dietary Supplement: Annona muricata

INTERVENTIONS:
Dietary Supplement: Annona muricata — Patients with prehypertension or stage 1 hypertension, in dietary measures, will received daily one tablet of 796 mg of aqueous extracts of Annona muricata leaves. During 60 days

SUMMARY:
The AM-HTN trial aim to investigate the effects of a tablet based on aqueous extracts of Annona muricata as add-on therapy in a hypertensive population.

Patients with prehypertension or stage 1 hypertension confirmed, will be selected and assign in a single arm, non randomly, open label clinical trial.

The group will receive in addition to their dietary measures, daily, one tablet of 796 mg of aqueous extracts of Annona muricata leaves.

The objective of AM-HTN is to determine the antihypertensive and metabolic effects of AM tablets in a population of African hypertensives.

Blood pressure profile, lipid profile, serum creatinine and transaminases profiles will be recorded and analysed at baseline and two months following enrolment.

DETAILED DESCRIPTION:
The AM-HTN trial aim to investigate the effects of a tablet based on aqueous extracts of Annona muricata as add-on therapy in a hypertensive population.

Patients with prehypertension or stage 1 hypertension confirmed, will be selected and assign in a single arm, non randomly, open label clinical trial.

The group will receive in addition to their dietary measures, daily, one tablet of 796 mg of aqueous extracts of Annona muricata leaves.

The objective of AM-HTN is to determine the antihypertensive and metabolic effects of AM tablets in a population of African hypertensives.

Blood pressure profile, lipids profile, serum creatinine and transaminases profiles were will be recorded and analysed at baseline and two months following enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure between 130/85 mmHg and 159/99 mmHg
* No antihypertensive therapy (determined by the investigator), except the hygiene dietetic measures, for at least 3 months
* No history of hepatic or renal insufficiency
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Side effects affecting life quality of patients (determined by the Data Safety and Monitoring Board).
* Out of sight.
* Withdrawal of consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Variation of the 24-hour systolic blood pressure (mmHg) | 60 days
  Variation of the 24-hour systolic blood pressure adjusted for baseline by using Ambulatory Blood Pressure Monitoring (ABPM)

SECONDARY OUTCOMES:
Variation in diurnal and nocturnal blood pressure (mmHg) | 60 days
  Variation of diurnal and nocturnal blood pressure profile adjusted for baseline by using ABPM
Variation in lipids profile (Triglycerides, HDL-cholesterol, LDL-cholesterol, Total cholesterol) on g/L | 60 days
  Variation on serum lipids (Triglycerides, HDL-cholesterol, LDL-cholesterol, Total cholesterol) profiles on g/L, adjusted for baseline. By Trinder Method on spectrophotometry.
Variation on serum creatinine (mg/L) and transaminases (SGOT/SGPT) profiles (UI/L) | 60 days
  Variation on serum creatinine (mg/L) by Jaffé Method and serum transaminases (SGOT/SGPT) profiles (UI/L)adjusted from baseline. By spectrophotometer.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nadege NGANOU-GNINDJIO, MD, MAS, Principal Investigator — Yaounde Central Hospital
Locations (1):
- Yaounde Central Hospital, Cardiology department, Yaoundé, Cameroon